CLINICAL TRIAL: NCT05996952
Title: A Multicenter Phase II Study of RC48-ADC in Adjuvant/Salvage Treatment of HER2 Positive High-risk Non-muscle-invasive Bladder Cancer
Brief Title: RC48-ADC in Adjuvant/Salvage Treatment of HER2 Positive Non-muscle-invasive Bladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hao Zeng, Professor, West China Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023(24)
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adjuvant RC48-ADC (Experimental): In this arm, RC48-ADC is evaluated in patients with HER2-positive high-risk non-muscle-invasive bladder cancer as an adjuvant treatment.
  Interventions: Drug: RC48-ADC
- Salvage RC48-ADC (Experimental): In this arm, RC48-ADC is evaluated in patients with HER2-positive non-muscle-invasive bladder cancer who failed BCG treatment as an adjuvant treatment.
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — Patients are treated with RC48-ADC at 2.0 mg/kg as an intravenous infusion over 30-90 minutes (60 minutes is recommended) once every 2 weeks for 12 weeks.

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC in adjuvant/salvage treatment of HER2 positive high-risk non-muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
This study is a multicenter phase II study, which aims to evaluate the efficacy and safety of intravenous RC48-ADC in adjuvant/salvage treatment of HER2 positive high-risk non-muscle-invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Life expectancy ≥12 weeks.
* Have a histologically-confirmed diagnosis of high-risk non-muscle-invasive (according to 2023 NCCN guidelines for bladder cancer) transitional cell carcinoma of the bladder. Subjects with tumors of mixed transitional/non-transitional cell histology are allowed, but transitional cell carcinoma must be the predominant histology.
* Have been treated with adequate BCG therapy and failed (according to 2023 EAU guidelines for NMIBC, for salvage treatment arm).
* Have elected not to undergo, or are considered ineligible for radical cystectomy, as determined by the treating surgeon.
* Have tumor tissues for HER2 IHC evaluation and have a HER2 expression score of HER2 2+ or HER2 3+ reviewed by an independent pathologist at the central laboratory.
* Have a performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Demonstrate adequate organ function.
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication.
* Male subjects of childbearing potential (Section 5.7.2) must agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy.

Exclusion Criteria:

* Has muscle-invasive (i.e. T2, T3, T4) locally advanced non-resectable or metastatic urothelial carcinoma.
* Has concurrent extra-vesical (i.e. urethra, ureter or renal pelvis) non-muscle invasive transitional cell carcinoma of the urothelium.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has undergone any intervening intravesical chemotherapy or immunotherapy from the time of most recent cystoscopy/TURBT to starting trial treatment. (Note: A single dose of intravesical treatment given as part of the most recent cystoscopy/TURBT, during the screening period, such as with chemotherapy as per local / regional practices, is acceptable.).
* Allergic to study therapy.
* Has a known additional malignancy that has had progression or has required active treatment in the last five years.
* Has an active autoimmune disease that has required systemic treatment in past 2 years.
* Have diseases that may interfere with the study treatment or severe and uncontrolled concomitant diseases.
* Has had an allogeneic tissue/solid organ transplant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
12-month recurence-free survival rate | From treatment initiation to 12 month
  The probability of patients remaining free of high-risk NMIBC or worse for at least 12 months after first dose of RC48-ADC adjuvant treatment
3-month pathological complete response rate | From treatment initiation to 3 month
  The proportion of patients are negative for urine cytology and cystoscopy at 3 month after first dose of RC48-ADC salvage treatment
Adverse events | From patient screening to 30 days after end of cycle 6
  The type, incidence, relatedness, and severity of adverse events

SECONDARY OUTCOMES:
6-month recurence-free survival rate | From treatment initiation to 6 month
  The probability of patients remaining free of high-risk NMIBC or worse for at least 6 months after first dose of RC48-ADC adjuvant treatment
Duration of response | From time of complete response to up to 60 months
  Time from complete response to recurrence of any disease
Recurrence-free survival | From time of first dose of RC48-ADC adjuvant treatment to up to 60 months
  Time from first dose of RC48-ADC adjuvant treatment to high-risk NMIBC recurrence or worse
Progression-free survival | From time of first dose of RC48-ADC treatment to up to 60 months
  Time from first dose of RC48-ADC treatment to progression to higher stage or death
Overall survival | From time of first dose of RC48-ADC treatment to up to 60 months
  Time from first dose of RC48-ADC treatment to death from any cause
Quality of life assessed by EQ-5D scale | After every cycle of treatment and 30 days after end of cycle 6
  Assessed by eEuroQoL EQ-5D scale, higher scores mean better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Hao Zeng, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No